CLINICAL TRIAL: NCT03746288
Title: A Multicenter, Randomized, Open-label, Controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of CAN008 Combined With Re-irradiation (rRT) for Treating Patients With Recurrent Glioblastoma (GBM)
Brief Title: To Evaluate the Efficacy and Safety of CAN008 Combined With Re-irradiation (rRT) for Treating Patients With Recurrent Glioblastoma (GBM)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CANbridge Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAN-B1-008-L-005
Record Dates: First submitted 2018-11-07; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: GBM
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): CAN008 400 mg weekly over no less than 30 minutes via intravenous drip, followed by rRT that same day
  Interventions: Drug: CAN008
- Control Group (Active Comparator): The dose is 2.0 Gy/d, 5 times/week, with a total planned radiation dose of 36 Gy.
  Interventions: Drug: CAN008

INTERVENTIONS:
Drug: CAN008 — CAN008 400 mg weekly over no less than 30 minutes via intravenous drip, followed by rRT that same day
  Other Names: Radiation

SUMMARY:
This is a multicenter, randomized, controlled study, aiming to evaluate the efficacy and safety of CAN008 administered once-weekly with rRT for treating first tumor recurrence in patients with GBM.

DETAILED DESCRIPTION:
This is a multi-center, randomized, controlled clinical trial to evaluate the efficacy and safety of CAN008 administered once-weekly with re-radiation therapy (rRT) in patients with an initial relapse of GBM. The subjects will be randomized into the treatment group (CAN008 + rRT) or the control group (rRT). The investigational treatment can be continued as long as the subjects have experienced lasting clinical benefits (complete response [CR], partial response [PR] or stable disease [SD]).

This study will be carried out in GBM subjects with an initial or second relapse. The subjects must have received standard care, including combination of radiotherapy and TMZ after surgical resection, and must be candidates for re-radiation therapy (rRT).

ELIGIBILITY:
Primary Inclusion Criteria:

1. Subjects with histologically diagnosed GBM confirmed by pathological tests at the central laboratory;
2. Subjects who have definite CD95L IHC expression level and CD95L methylation level results confirmed at the central laboratory;
3. Subjects with GBM who are not suitable for surgical ablation after tumor recurrence or have residual neoplasm after surgical ablation;
4. Patients with disease progression or recurrence based on RANO (Response Assessment in Neuro-oncology) Criteria identified upon magnetic resonance imaging (MRI) performed two weeks prior to the first dose of investigational drug and two weeks prior to the initiation of rRT;
5. Age ≥ 18 years and ≤ 70 years;
6. Expected survival ≥ 3 months;
7. Karnofsky score ≥60;
8. Subjects who have tumor progression after having previously received standard treatments including surgery, chemoradiation combination (RT+ TMZ), adjuvant chemotherapy (TMZ);
9. Subjects who have a single primary lesion or have scattered or multiple lesions which can be contained within a radiation target volume;
10. Subjects who have received a maximum dose of 60 Gy for a single tumor in situ in the previous RT, or have not received RT for at least 8 months;
11. Subjects eligible to receive rRT who have recurrence of tumor in situ on the T1-weighted MRI (T1-MRI) (Gd), with the maximum diameter of 1-4 cm;
12. Subjects who have appropriate hematologic parameters (absolute neutrophil count (ANC) ≥1.5×109/L, platelet count ≥80×109/L, hemoglobin (Hb)≥90 g/L), kidney function (serum creatinine≤1.25×ULN) and liver function (total bilirubin≤1. 5×ULN, AST≤2.5×ULN and ALT≤2.5×ULN);
13. Subjects treated with hormone therapy must receive the treatment with steroid hormones at a stable dose or a reduced dose within 5 days before entering the trial;
14. Female subjects of childbearing potential must have a negative serum HCG pregnancy test within 7 days before the first dose of investigational drug;
15. Male and female subjects of childbearing potential must agree to adopt approved contraceptive methods (such as condoms and intrauterine ring) during the trial and till 3 months after the completion of this trial;
16. Subjects who are willing and able to comply with regulations specified in the clinical trial protocol (as judged by investigators);
17. Subjects who have signed the Informed Consent Form (ICF);

Primary Exclusion Criteria:

1. Subjects who have previously received more than one course of RT for the head or have received a total dose of >60 Gy in the previous RT;
2. Subjects who have received an accumulated radiation dose of >54 Gy for the optic chiasma;
3. Subjects whose scattered or multiple tumors cannot be included within a radiation target volume;
4. Subjects who have previously received treatment with bevacizumab, iodine radiotherapy, gamma knife and/or brachytherapy;
5. Subjects who cannot undergo MRI examination or follow-ups;
6. Subjects with human immunodeficiency virus (HIV) infection;
7. Subjects with active viral hepatitis need to be excluded:

   * For those with inactive viral hepatitis, they can be considered to be enrolled in this trial if their liver function is within the allowable range, that is, hepatitis B virus deoxyribonucleic acid (HBV- DNA)<2,000 IU/Ml;
   * For those infected with hepatitis C virus (HCV), they can also be considered to be included if no HCV ribonucleic acid (HCV-RNA) is detected;
8. Subjects who have hereditary fructose intolerance (HFI);
9. Subjects whose previous history (such as serious coronary heart disease, serious diabetes, immune deficiency, sequelae of apoplexia, serious mental retardation, etc.) is considered to indicate poor prognosis, as evaluated by investigators;
10. Pregnant and breast-feeding women;
11. Subjects who suffer from any malignant tumors (except for basal cell carcinoma or cervical carcinoma in situ) at the same time. Those who have previously suffered from malignant tumors but have no evidences of disease recurrence for at least 5 years can still participate in this trial;
12. Subjects who have participated in other clinical trials within 30 days prior to the enrollment or during the treatment phase of this trial;
13. Subjects who has known coronary heart disease complicated by serious cardiac arrhythmias or heart failure (NYHA III-IV).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause,assessed up to 12 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | "From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
6-month progression free survival rate (PFS6) | The percentage of subjects confirmed without PD or death at 6 months after randomization.
Objective response rate (ORR) | rom date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 8 months").
Duration of response (DOR) | rom date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 8 months").

IPD SHARING:
Plan to Share IPD: No